CLINICAL TRIAL: NCT05079568
Title: "A Pilot Study to Assess the Safety, Tolerability and Efficacy of Virtual Reality for the Treatment of Gastroparesis"
Brief Title: A Study to Evaluate the Safety and Tolerability of Virtual Reality to Treat Gastroparesis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Lacy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-007072
Record Dates: First submitted 2021-10-02; First posted 2021-10-15 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind, randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active VR Group (Experimental): Subjects will be provided an Oculus Go VR headset pre-loaded with a "menu" of virtual reality programs which have been designed specifically to treat both acute and chronic pain. Subjects are required to use the VR headset at home four times daily, prior to breakfast, lunch, dinner, and bedtime. Each session will last approximately 15 minutes.
  Interventions: Device: Oculus Go VR headset
- Sham VR Group (Sham Comparator): Subjects will be provided an Oculus Go VR headset pre-loaded two-dimensional nature video. Subjects are required to use the VR headset at home four times daily, prior to breakfast, lunch, dinner, and bedtime. Each session will last approximately 15 minutes.
  Interventions: Device: Sham Oculus Go VR headset

INTERVENTIONS:
Device: Oculus Go VR headset — Virtual reality programs consisting of interactive games, meditation and deep breathing exercises, and passive virtual reality experiences designed to facilitate relaxation.
  Arms: Active VR Group
Device: Sham Oculus Go VR headset — Virtual reality program with two-dimensional nature video
  Arms: Sham VR Group

SUMMARY:
The purpose of this study is to determine if virtual reality therapy is safe and tolerable in treating gastroparesis.

DETAILED DESCRIPTION:
After informed consent patients will be randomized to a 4 week treatment program comparing active VR treatment to sham VR treatment. Symptoms will be measured at baseline and at 2 and 4 weeks using validated questionnaires. A short questionnaire will be answered daily to evaluate changes in nausea.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, men and women ages 18-75.
* Documented gastroparesis (idiopathic or diabetic).
* Patients who have had an upper endoscopy within the past 3 years not showing evidence of an organic disorder that could cause symptoms and a 4-hour scintigraphic gastric emptying scan showing evidence of delayed gastric emptying.
* Patients will be identified as direct referrals to the general GI clinic or the motility clinic, and will undergo screening history and physical examination by the PI or co-investigator.

Exclusion Criteria:

* Patients whose symptoms are thought to represent an organic disorder (e.g., peptic ulcer disease, hepatitis, pancreatitis, inflammatory bowel disease, a known malignancy, radiation-induced injury, an active infection, vasculitis, celiac disease).
* If the patients have known uncontrolled diabetes (HgbA1c > 11), GERD, esophagitis, eosinophilic esophagitis, H. pylori, cannabinoid hyperemesis syndrome, celiac artery compression syndrome, or SMA syndrome.
* Patients with prior surgery to the esophagus, stomach or duodenum.
* Patients taking opioids will also be excluded.
* Alcohol and tobacco use will be assessed, as will the presence of psychiatric conditions, such as anxiety, depression, post-traumatic stress disorder, bipolar disorders, and eating disorders, such as anorexia nervosa and bulimia. However, no patient will be excluded based on reported substance use or presence of a psychiatric comorbidity, unless their psychological status represents potential harm to themselves, others, or represents an impediment to treatment.
* Any patient identified as having a significant problem with alcohol or anxiety or depression will be referred back to their primary care provider for further evaluation and treatment.
* Patients with motion sickness, vertigo, or a seizure disorder will be excluded to prevent the theoretical risk of inducing or exacerbating symptoms related to the aforementioned conditions with VR.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported adverse events | 4 weeks
  Number of patient-reported adverse events assessed using standardized daily patient-reported adverse event questionnaires

SECONDARY OUTCOMES:
Changes in global gastroparesis symptom scores | Baseline, 4 weeks
  Measured by the self-reported GCSI (Gastroparesis Cardinal Symptom Index-daily diary); consisting of questions about severity of symptoms experienced during the past 24 hours on a scale of none, mild, moderate, severe, and very severe.
Changes in gastrointestinal disorder symptoms | Baseline, 4 weeks
  Measured using the Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) questionnaire; consisting of questions about severity of symptoms related to gastrointestinal problem during the past 2 weeks on a scale of 0=note to 5=very severe.
Changes in individual scores for nausea | Baseline, 4 weeks
  Measured using Visual Analogue Scale (VAS) where subject place a X on a scale to show how much nausea they had today; scale is 0%=no nausea, 100%=worse nausea ever.
Changes in abdominal pain | Baseline, 4 weeks
  Measured using a Numeric Pain Rating Scale (NRS) where subject place a X on a scale to show how much abdominal pain they had today; scale is 0% no abdominal pain, 100% worse abdominal pain ever.
Changes in bloating | Baseline, 4 weeks
  Measured using the validated Mayo Bloating Questionnaire to assess subject symptoms of gastroparesis
Change in work productivity | Baseline, 4 weeks
  Measured using the validated WPAI (work productivity activity index) to assess subject ability to work and perform regular activities
Change in Quality of life | Baseline, 4 weeks
  Measured using the self-reported Short-Form 12 questionnaire; health survey to assess subject views about their health

CONTACTS AND LOCATIONS:
Overall Officials: Brian Lacy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials